CLINICAL TRIAL: NCT04571307
Title: Pilot Study on the Feasibility of Cryotherapy as an Alternative Treatment for Phyllodes Tumors/Breast Fibroepithelial Lesions (FELs) Needing Surgery
Brief Title: Cryotherapy in Breast B3 Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019/2944
Record Dates: First submitted 2020-08-31; First posted 2020-10-01 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Breast Disease; Phyllodes Breast Tumor
MeSH Terms: conditions — Breast Diseases; Phyllodes Tumor | interventions — Cryotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cryotherapy — comparison between cryotherapy and surgery

SUMMARY:
To determine the feasibility of cryotherapy for B3 fibroepithelial lesions

ELIGIBILITY:
Inclusion Criteria:

* lesion seen on ultrasound
* core biopsy revealed FEL of B3
* lesion </+3.5cm
* keen for cryotherapy instead of surgery
* has other breast lesions for followup

Exclusion Criteria:

* cancer patients
* patients with bleeding diathesis
* lesions causing visible breast deformity

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
recurrence of the lesion | 2 years from procedure
  assessed on ultrasound
breast cosmetic outcome | at 1 year post procedure
  patient self assessment of excellent (1), good (2), fair (3) poor (4). score of 1-4,1 being the best score
pain score | immediate post procedure
  using pain score scale of 0-10, a higher score indicates a worse outcome
pain score | at 2 weeks post procedure
  using pain score scale of 0-10, a higher score indicates a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Geok hoon lim, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore